CLINICAL TRIAL: NCT02305524
Title: Evaluation of Chest Compression Effect on Airway Management With he Visualized Tracheoscopic Ventilation Tube and the Macintosh Laryngoscopy by Novice Paramedics: a Randomized Crossover Simulation Study.
Brief Title: Intubation During Adult Intubation
Acronym: SLETI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Institute of Rescue Research and Education (Other)
Responsible Party: Principal Investigator, Lukasz Szarpak, Lukasz Szarpak, National Institute of Cardiology, Warsaw, Poland
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ETI/2014/44
Record Dates: First submitted 2014-11-27; First posted 2014-12-02 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Cardiac Arrest
Keywords: endotracheal intubation
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ETI with chest compressions (Experimental): endotracheal intubation (ETI) during child mannikin resuscitation with uninterrupted chest compressions. In order to simulate the difficulties associated with intubation during uninterrupted chest compressions, CPR was performed by using LUCAS-2 (Physio-Control, Redmond, WA, U.S.).
  Interventions: Device: ETView VivaSight SL; Device: Macintosh laryngoscope
- ETI without chest compressions (Experimental): Endotracheal intubation of child mannikin during resuscitation without chest compressions.
  Interventions: Device: ETView VivaSight SL; Device: Macintosh laryngoscope

INTERVENTIONS:
Device: ETView VivaSight SL — Intubation using ETView VivaSight SL
Device: Macintosh laryngoscope — intubation with macintosh laryngoscope with conventional tube

SUMMARY:
The objective of this study is to compared effectiveness of intubation using ETView VivaSight SL and standard tracheal tube during resuscitation performed by a EMS-paramedics.

ELIGIBILITY:
Inclusion Criteria:

* Give voluntary consent to participate in the study
* minimum 1 year of work experience in emergency medicine
* experienced emergency medical personnel (physicians, nurses, paramedics)

Exclusion Criteria:

* Not meet the above criteria
* Wrist or Low back diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-11; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Success of intubation | 1 day
  effectiveness of the first, second and third intubation attempts and overall effectiveness of intubation by participants using four intubation devices. If the examinee failed at all attempts, the case was excluded from the time calculations.

SECONDARY OUTCOMES:
Time to intubation | 1 day
  time from insertion of the blade to the first manual ventilation of the manikin´s lungs. If time of intubation is over than 60 seconds, attempt was recognized as failure.
Cormack-Lehan scale | 1 day
  self reported Cormack-Lehan scale during intubation

CONTACTS AND LOCATIONS:
Locations (1):
- International Institute of Rescue Research and Education, Warsaw, Masovia, Poland